CLINICAL TRIAL: NCT00792389
Title: Randomised Controlled Trail of Warmed Humidified Insufflation Versus Cold Non-Humidified Insufflation in Elective Laparoscopic Cholecystectomies: Does This Reduce Post-Operative Pain?
Brief Title: Study of the Use of Humidified Warmed Gas and the Effect on Post-Operative Pain in Laparoscopic Cholecystectomies
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Pennine Acute Hospitals NHS Trust (Other)
Responsible Party: Mr David Flook, Pennine Acute NHS Hospitals Trust
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PAT-HWA-001
Record Dates: First submitted 2008-11-14; First posted 2008-11-17 (Estimated); Last update posted 2008-11-17 (Estimated); Status verified 2008-11

CONDITIONS: Gallstone
Keywords: Gallstones; Gallbladder; Cholecystectomy; Gallstone disease
MeSH Terms: conditions — Gallstones; Cholelithiasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Patients receiving warmed, humidified gas
  Interventions: Other: Warm humidified C02
- 2 (Active Comparator): Patients receiving cool, day gas
  Interventions: Other: Cool dry C02

INTERVENTIONS:
Other: Warm humidified C02 — Insufflation of warmed humidified gas during laparoscopic cholecystectomy
  Other Names: Fisher Paykall laparoscopic humidifier
  Arms: 1
Other: Cool dry C02 — Insufflation of cool dry gas during laparoscopic cholecystectomy
  Arms: 2

SUMMARY:
Double blind RCT comparing elective laparoscopic cholecystectomy using warmed, humidified gas (new) against laparoscopic cholecystectomy with cool, dry gas (usual). Sample size of 200 patients. Outcome measures are postoperative opiate analgesia use, and post operative numerical pain scores.

ELIGIBILITY:
Inclusion Criteria:

* elective laparoscopic cholecystectomy
* 18 years of age or over

Exclusion Criteria:

* under 18 years of age
* prisoners
* converted to open operation
* secondary invasive procedure during operation
* unable to give consent for whatever reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-01 (Estimated); Study Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
Total post operative opiate analgesia - morphine equivalent dose. | 1 day

SECONDARY OUTCOMES:
Subjective post operative pain as defined on numerical pain scales | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: David Flook, MBChB, Principal Investigator — Pennine Acute Hospital NHS Trust
Locations (1):
- Royal Oldham Hospital, Oldham, Lancashire, United Kingdom